CLINICAL TRIAL: NCT00292981
Title: Open-label Extension Study of CE1145 (Human Pasteurized C1 Esterase Inhibitor Concentrate) in Subjects With Congenital C1-INH Deficiency and Acute HAE Attacks
Brief Title: C1 Esterase Inhibitor in Hereditary Angioedema (HAE)(Extension Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE1145_3003; 1453 (Other: CSL Behring)
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2011-10

CONDITIONS: Hereditary Angioedema
Keywords: C1 Inhibitor; Hereditary angioedema; Acute HAE attack
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

ARMS (1):
- C1 Esterase Inhibitor (Experimental)
  Interventions: Drug: C1 Esterase Inhibitor

INTERVENTIONS:
Drug: C1 Esterase Inhibitor — Lyophilisate containing approximately 500 U C1-INH to be reconstituted with 10 mL water for injection; Single Dose: 20 U/kg b.w. iv
  Other Names: Berinert P

SUMMARY:
Hereditary angioedema (HAE) is a rare disorder characterized by congenital lack of functional C1 esterase inhibitor. If not treated adequately, the acute attacks of HAE can be life-threatening and may even result in fatalities, especially in case of involvement of the larynx.The planned extension study is designed to enrol subjects that participated in the pivotal study in order to provide them with C1-INH for treatment of acute HAE attacks for 24 months or until the licensing procedure for C1-INH is finalized, whatever comes first.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented congenital C1-INH deficiency
* Acute HAE attack
* Participation in base study CE1145_3001 (NCT00168103)

Key Exclusion Criteria:

* Acquired angioedema
* Treatment with any other investigational drug besides CE1145 in the last 30 days before study entry

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-08; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (14):
- United States (13):
  - Contact CSL Behring for facility details, Weston, Florida
  - Contact CSL Behring for facility details, Atlanta, Georgia
  - Contact CSL Behring for facility details, Idaho Falls, Idaho
  - Contact CSL Behring for facility details, Chicago, Illinois
  - Contact CSL Behring for facility details, Shreveport, Louisiana
  - Contact CSL Behring for facility details, Boston, Massachusetts
  - Contact CSL Behring for facility details, Plymouth, Minnesota
  - Contact CSL Behring for facility details, Omaha, Nebraska
  - Contact CSL Behring for facility details, Tulsa, Oklahoma
  - Contact CSL Behring for facility details, Eugene, Oregon
  - Contact CSL Behring for facility details, Hershey, Pennsylvania
  - Contact CSL Behring for facility details, Rapid City, South Dakota
  - Contact CSL Behring for facility details, Dallas, Texas
- Contact CSL Behring for facility details, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Craig TJ, Wasserman RL, Levy RJ, Bewtra AK, Schneider L, Packer F, Yang WH, Keinecke HO, Kiessling PC. Prospective study of rapid relief provided by C1 esterase inhibitor in emergency treatment of acute laryngeal attacks in hereditary angioedema. J Clin Immunol. 2010 Nov;30(6):823-9. doi: 10.1007/s10875-010-9442-1. Epub 2010 Jul 16. PMID 20635155
- [Background] Bernstein JA, Machnig T, Keinecke HO, Whelan GJ, Craig TJ. The effect of weight on the efficacy and safety of C1 esterase inhibitor concentrate for the treatment of acute hereditary angioedema. Clin Ther. 2014 Apr 1;36(4):518-25. doi: 10.1016/j.clinthera.2014.02.005. Epub 2014 Mar 21. PMID 24661784
- [Background] Bork K, Craig TJ, Bernstein JA, Feuersenger H, Machnig T, Staubach P. Efficacy of C1 esterase inhibitor concentrate in treatment of cutaneous attacks of hereditary angioedema. Allergy Asthma Proc. 2015 May-Jun;36(3):218-24. doi: 10.2500/aap.2015.36.3844. Epub 2015 Mar 23. PMID 25803207
- [Result] Wasserman RL, Levy RJ, Bewtra AK, Hurewitz D, Craig TJ, Kiessling PC, Keinecke HO, Bernstein JA. Prospective study of C1 esterase inhibitor in the treatment of successive acute abdominal and facial hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2011 Jan;106(1):62-8. doi: 10.1016/j.anai.2010.10.012. Epub 2010 Nov 20. PMID 21195947
- [Result] Craig TJ, Bewtra AK, Bahna SL, Hurewitz D, Schneider LC, Levy RJ, Moy JN, Offenberger J, Jacobson KW, Yang WH, Eidelman F, Janss G, Packer FR, Rojavin MA, Machnig T, Keinecke HO, Wasserman RL. C1 esterase inhibitor concentrate in 1085 Hereditary Angioedema attacks--final results of the I.M.P.A.C.T.2 study. Allergy. 2011 Dec;66(12):1604-11. doi: 10.1111/j.1398-9995.2011.02702.x. Epub 2011 Sep 2. PMID 21884533
- [Derived] Craig TJ, Rojavin MA, Machnig T, Keinecke HO, Bernstein JA. Effect of time to treatment on response to C1 esterase inhibitor concentrate for hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2013 Sep;111(3):211-5. doi: 10.1016/j.anai.2013.06.021. Epub 2013 Jul 16. PMID 23987198
- [Derived] Craig TJ, Bewtra AK, Hurewitz D, Levy R, Janss G, Jacobson KW, Packer F, Bernstein JA, Rojavin MA, Machnig T, Keinecke HO, Wasserman RL. Treatment response after repeated administration of C1 esterase inhibitor for successive acute hereditary angioedema attacks. Allergy Asthma Proc. 2012 Jul-Aug;33(4):354-61. doi: 10.2500/aap.2012.33.3589. PMID 22856636
- See also: United States Hereditary Angioedema Association — http://www.hereditaryangioedema.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, open-label extension study enrolling subjects at 15 sites in North America that had participated in study CE1145_3001 (NCT00168103). Enrollment occurred between August 2005 and January 2008.
Period: Overall Study
Arm/Group | C1 Esterase Inhibitor
Started | 57
Completed | 18
Not Completed | 39
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 13
Not completed — Withdrawal by Subject | 22
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 19
Type of HAE [Number; unit: participants] — Type I HAE (common form genotype): An impaired synthesis and an elevated turnover of a normal and functionally active C1-Inhibitor (C1-INH) molecule occurs, causing a reduction in the availability of functionally active C1-INH to levels of 5% to 30% of normal.
  Type II HAE (variant form genotype): Normal levels of a functionally impaired C1-INH molecule are synthesized while the normal form of C1-INH is considerably reduced in the circulation.
  participants
    Type I HAE | 49
    Type II HAE | 7
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Start of Relief of Symptoms From HAE Attack (Intent to Treat (ITT) Subject Population)
Description: The start of symptom relief was determined by subject self-assessment.
Time Frame: Up to 24 h after start of study treatment
Population: Intent to treat (ITT) subject population: All subjects admitted to the study who received any portion of the study medication.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 57
hours | 0.46 [0.39 to 0.53]

2. Secondary Outcome: Time to Complete Resolution of All HAE Symptoms (ITT Subject Population)
Description: Complete resolution of symptoms was determined by subject self-assessment and documented on a diary card.
Time Frame: Up to Day 9 following an attack
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 57
hours | 15.48 [11.64 to 21.59]

3. Primary Outcome: Time to Start of Relief of Symptoms From HAE Attack (ITT Attack Population)
Description: The start of symptom relief was determined by subject self-assessment.
Time Frame: Up to 24 h after start of study treatment
Population: ITT attack population: All attacks in subjects admitted to the study for which any portion of study medication was administered.
Measure: Median (95% Confidence Interval); unit: hours
Units Other Than Participants: HAE Attacks
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 57
Number analyzed (HAE Attacks) | 1085
hours | 0.37 [0.33 to 0.42]

4. Secondary Outcome: Time to Complete Resolution of All HAE Symptoms (ITT Attack Population)
Description: Complete resolution of symptoms was determined by subject self-assessment and documented on a diary card.
Time Frame: Up to Day 9 following an attack
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: hours
Units Other Than Participants: HAE Attacks
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 57
Number analyzed (HAE Attacks) | 1085
hours | 14.28 [12.07 to 15.80]

ADVERSE EVENTS:
Time Frame: For each HAE attack, the AE reporting period comprised the time period from the subject's enrollment (Day 1) until Day 7 to 9. The reporting period for serious adverse events (SAEs) was 12 Weeks from the time of the first HAE attack.
Description: Adverse events were documented in a diary card. Subjects were treated for 1 to 186 attacks during the study. The safety population consisted of enrolled subjects who received study medication.
Arm/Group | C1 Esterase Inhibitor
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 25/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C1 Esterase Inhibitor (N=57)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 — A hereditary angioedema attack was reported as an adverse event if it represented a worsening of symptoms during a treated attack.
Staphylococcal infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C1 Esterase Inhibitor (N=57)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 — A hereditary angioedema attack was reported as an adverse event if it represented a worsening of symptoms during a treated attack.
Conjunctivitis (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 2
Local swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Infusion related reaction (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2
Erythema infectiosum (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Periodontal infection (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Vaginitis bacterial (Infections and infestations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Blood potassium decreased (Investigations) | 1
Red blood cells urine positive (Investigations) | 1
Urine leukocyte esterase positive (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned before seeking publication review.